CLINICAL TRIAL: NCT07325617
Title: The TALK-U Study: Tracking AI/LLM Knowledge and Use in Urology Outpatients and Its Association With Anxiety, Satisfaction, and Health Awareness-A Cross-Sectional Study
Brief Title: Tracking AI/LLM Literacy and Knowledge in Urology Outpatients (TALK-U)
Acronym: TALK-U
Status: Not yet recruiting | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Tuncel Uzel, Principal Investigator, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: 2025-06/98
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Health Information Seeking Behavior; Anxiety
Keywords: Artificial intelligence; Anxiety; ChatGPT; Gemini; Health information seeking; Large language model (LLM); Patient satisfaction
MeSH Terms: conditions — Anxiety Disorders; Patient Satisfaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AI/LLM users: Participants who report prior use of AI chat tools based on large language models (e.g., ChatGPT or similar) for health information before the outpatient urology visit, as assessed by the study questionnaire.
- non AI/LLM users: Participants who report no prior use of AI/LLM chat tools (e.g., ChatGPT or similar) for health information before the outpatient urology visit, as assessed by the study questionnaire.

SUMMARY:
This study is a one-time, questionnaire-based survey of adults attending a urology outpatient clinic. The investigators will examine whether patients who use AI chat tools based on large language models (LLMs), such as ChatGPT, before seeking care differ from non-users in (1) anxiety, (2) satisfaction with the clinic visit, and (3) awareness/understanding of their health condition.

Participants who provide written informed consent will complete a brief survey during their clinic visit (about 5-7 minutes). The survey includes a standardized anxiety scale (GAD-7), visual analog scales (0-10) for anxiety before and after the visit, satisfaction, and disease awareness, as well as questions about AI/LLM knowledge and use. Treating clinicians will not have access to participants' survey responses, and participation will not affect clinical care.

DETAILED DESCRIPTION:
The TALK-U study is a cross-sectional, observational survey conducted in the urology outpatient clinic of Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital. The primary exposure is self-reported AI/LLM knowledge and use for health information (e.g., whether participants have used ChatGPT or similar tools, frequency, awareness of AI, and purpose of use). The primary outcome is anxiety measured by GAD-7 at the time of the clinic encounter. Secondary outcomes include (i) anxiety assessed on a 0-10 visual analog scale before and after the visit, (ii) outpatient visit satisfaction (0-10 VAS), and (iii) perceived disease awareness/understanding (0-10 VAS).

Eligible adult first-time urology outpatients who can complete the survey independently and provide informed consent will be invited during a 2-month recruitment period. Analyses will compare outcomes between AI/LLM users and non-users and explore associations with age group (<40, 40-60, >60), education level, and urology subspecialty category. Data will be analyzed using appropriate parametric/nonparametric tests depending on distribution, with p < 0.05 considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* First-time visit to the Urology Outpatient Clinic
* Able to read and write and complete the questionnaire independently
* Able to provide written informed consent

Exclusion Criteria:

* Age under 18 years
* Insufficient literacy to understand and complete the questionnaire
* Severe hearing or visual impairment, or a neurological/psychiatric condition that prevents understanding and completing the survey
* Refusal or inability to provide informed consent
* Currently under follow-up for a known urologic condition (i.e., not a first-time urology outpatient visit)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) presenting for a first-time visit to the Urology Outpatient Clinic at Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital will be invited to participate during a 2-month recruitment period. Participants who provide written informed consent and can complete a brief questionnaire independently will be enrolled. The study will include both sexes and a broad range of urologic presenting complaints.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Pre-visit Anxiety (VAS 0-10) | Day 0 (immediately before the outpatient visit)
  Self-rated anxiety on a 0-10 visual analog scale (VAS), where 0 indicates no anxiety and 10 indicates the highest possible anxiety. This measure reflects visit-related state anxiety prior to clinician encounter.

SECONDARY OUTCOMES:
Post-visit Anxiety (VAS 0-10) | Day 0 (immediately after the outpatient visit)
  Self-rated anxiety on a 0-10 VAS (0 = none, 10 = highest).
Visit Satisfaction (VAS 0-10) | Day 0 (immediately after the outpatient visit)
  Self-rated satisfaction with the outpatient visit on a 0-10 VAS (0 = not satisfied at all, 10 = maximum satisfaction).
Disease Awareness/Understanding (VAS 0-10) | Day 0 (during the outpatient clinic visit)
  Self-rated awareness/understanding of one's condition on a 0-10 VAS (0 = none, 10 = complete).

OTHER OUTCOMES:
Baseline General Anxiety Symptoms (GAD-7 Total Score) | Day 0 (at enrollment; prior to or during the clinic visit)
  Total score on the 7-item GAD-7 questionnaire (range 0-21; higher scores indicate greater generalized anxiety symptoms). This measure will be used to account for baseline anxiety (trait-like symptoms) and to adjust analyses of VAS-based state anxiety out

CONTACTS AND LOCATIONS:
Locations (1):
- Dr.Abdurrahman Yurtaslan Ankara Oncology Research and Training Hospital, Ankara, Yenimahalle/Ankara, Turkey (Türkiye)